CLINICAL TRIAL: NCT00532363
Title: Obesity-related Pseudo-asthma (ORPA): Description of a Novel Clinical Entity
Brief Title: Obesity and Asthma:a Specific Phenotype
Acronym: ORPA
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Louis-Philippe Boulet, MD, FRCPC, FCCP, Laval University
Other Study IDs: HL-ORPA-1171
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Obesity; Asthma
MeSH Terms: conditions — Obesity; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese asthmatics: Obese subjects with asthma (on inhaled corticosteroids)
- Non obese asthmatics: Non obese subjects with asthma (on inhaled corticosteroids)

SUMMARY:
Clinicians frequently observed that obese women referred for severe asthma do not respond to treatment. These patients, despite the presence of wheezing, often have normal expiratory flows and normal or "borderline" airway responsiveness.

It is therefore possible that this mode of presentation reflect a pseudo-asthmatic state for which clinical definition and characteristics and optimal management remain to be determined.

The aim of this study was to study the pulmonary physiological and airway inflammatory characteristics and response to treatment of obese women considered to have clinically severe asthma in order to demonstrate that some of these patients have a phenotype that is not that of asthma.

DETAILED DESCRIPTION:
Twenty-five obese women (BMI over 30) and 25 non-obese women (18>BMI<25) considered to have severe asthma by their physician and requiring corticosteroids to control their asthma will have the following investigation:

* Respiratory questionnaires focussing on the nature and time-course of symptoms, asthma control criteria, medication use.
* Physical examination, including measures of BMI, waist, hips and ratio waist/hips
* Blood test for Complete Blood Count, blood glucose, total IgE levels and markers of systemic inflammation (C-Reactive Protein, fibrinogen…)
* Spirometry and bronchodilator response.
* Induced sputum analysis and Exhaled Breath Condensate pH to assess airway inflammation.
* Skin prick tests with a battery of common airborne allergens
* Measurement of lung volumes and airway resistance + MIP and MEP.
* Methacholine challenge (up to 16 mg/ml) with Borg scores for breathlessness and chest tightness.

ELIGIBILITY:
Inclusion Criteria:

* Will be women aged 18 years and over
* Will be in good health apart from asthma or obesity as determined by history and physical examination (No other condition that could influence the proposed tests).
* All will be non smokers or ex-smokers for more than six months with a smoking history of no more than 10 pack- years (i.e., one pack per day or its equivalent for 10 years.)
* Subjects will have a physician's made diagnosis of severe asthma and treated with corticosteroids.

Exclusion Criteria:

* Subjects who are, in the opinion of the investigator, mentally or legally incapacitated thus preventing informed consent from being obtained.
* Subjects having a co-existing illness that precludes them from the trial.
* Pregnancy or lactation
* Contraindication to the prednisone treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from advertisements in newspapers and from the hospital primary care asthma clinic and will be offered to participate to the study.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2005-09; Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Hôpital Laval
Locations (1):
- Centre de Recherche, Hôpital Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Lessard A, Turcotte H, Cormier Y, Boulet LP. Obesity and asthma: a specific phenotype? Chest. 2008 Aug;134(2):317-323. doi: 10.1378/chest.07-2959. Epub 2008 Jul 18. PMID 18641097